CLINICAL TRIAL: NCT01066052
Title: Collaborative Study to Assess the Effects of Treatment With Recombinant Growth Hormone Saizen® in the Prevention of Short Stature in Young Girls Suffering From Turner Syndrome Before the Age of 4 Years. Original French Title: Etude Collaborative Pour apprécier Les Effets du Traitement Par l'Hormone de Croissance Recombinante SAIZEN® Dans le Retard de Croissance de la Fillette Atteinte de Syndrome de Turner Avant l'âge de 4 Ans
Brief Title: Growth Hormone Treatment for the Prevention of Short Stature in Young Girls With Turner Syndrome Before the Age of 4 Years
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GF 5834
Record Dates: First submitted 2010-02-05; First posted 2010-02-10 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-06

CONDITIONS: Turner's Syndrome
Keywords: Growth hormone; Turner syndrome; r-hGH; early treatment
MeSH Terms: conditions — Turner Syndrome | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- r-hGH (Experimental): Participants (girls) will receive r-hGH as a subcutaneous injection administered by a parent in the evening. During Years 1-2, the dose of r-hGH received will depend on participants' baseline height standard deviation score (SDS) relative to the general population standard: participants with a height SDS of -2 standard deviation (SD) or lower will receive 0.05 milligrams per kilogram (mg/kg) per day r-hGH and those with a height SDS between -1 and -2 SD will receive 0.035 mg/kg per day r-hGH. After 2 years of treatment, all participants will receive a fixed dose of 0.05 mg/kg per day for a further 2 years.
  Interventions: Drug: r-hGH
- Historical Control (No Intervention): This arm will include matching (age and height) historical control participants (girls) with turner syndrome, who were born between 1961 and 1990 and were untreated.

INTERVENTIONS:
Drug: r-hGH — Subcutaneous administration.
  Other Names: Saizen®
  Arms: r-hGH

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of recombinant human growth hormone (r-hGH) treatment in girls with Turner Syndrome under the age of 4 years. After 4 years of treatment, height in these girls will be compared with an historical control group of untreated girls with Turner Syndrome, matched for age and height at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Young girls with turner syndrome proved by karyotype
* Growth hormone secretion confirmed with ornithin stimulation test
* Normal glucidic metabolism confirmed by assessment of HbA1c
* None associated severe pathology which could have impact on growth (i.e. renal insufficiency, decompensated heart failure)
* No previous or associated treatment with anabolic or sexual steroids
* Known parental height

Exclusion Criteria:

* Severe associated pathology with impact on growth
* Concomitant treatment with impact on growth
* Previous or associated treatment with anabolic steroids
* Associated growth hormone deficiency

Max Age: 4 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 1992-02-29 (Actual); Primary Completion 1999-03-31 (Actual); Study Completion 2010-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- Hôpital Robert Debré, Paris, France

REFERENCES:
- [Result] Linglart A, Cabrol S, Berlier P, Stuckens C, Wagner K, de Kerdanet M, Limoni C, Carel JC, Chaussain JL; French Collaborative Young Turner Study Group. Growth hormone treatment before the age of 4 years prevents short stature in young girls with Turner syndrome. Eur J Endocrinol. 2011 Jun;164(6):891-7. doi: 10.1530/EJE-10-1048. Epub 2011 Mar 11. PMID 21398400

RESULTS

PARTICIPANT FLOW:
Groups:
- Recombinant Human Growth Hormone (r-hGH): Participants (girls) received r-hGH (Saizen®) as a subcutaneous injection administered by a parent in the evening. During Years 1-2, the dose of r-hGH received depended on participants' baseline height standard deviation score (SDS) relative to the general population standard: participants with a height SDS of -2 standard deviation (SD) or lower received 0.05 milligrams per kilogram (mg/kg) per day r-hGH and those with a height SDS between -1 and -2 SD received 0.035 mg/kg per day r-hGH. After 2 years of treatment, all participants received a fixed dose of 0.05 mg/kg per day for a further 2 years.
- Historical Control: This arm included matching (age and height) historical control participants (girls) with turner syndrome, who were born between 1961 and 1990 and were untreated.
Period: Overall Study
Arm/Group | Recombinant Human Growth Hormone (r-hGH) | Historical Control
Started | 64 | 51
Treated | 61 | 0
Completed | 61 | 51
Not Completed | 3 | 0
Not completed — Enrolled But Not Treated | 3 | 0

BASELINE CHARACTERISTICS:
Population: All Participants.
Groups:
- r-hGH: Participants (girls) received r-hGH as a subcutaneous injection administered by a parent in the evening. During Years 1-2, the dose of r-hGH received depended on participants' baseline height SDS relative to the general population standard: participants with a height SDS of -2 SD or lower received 0.05 mg/kg per day r-hGH and those with a height SDS between -1 and -2 SD received 0.035 mg/kg per day r-hGH. After 2 years of treatment, all participants received a fixed dose of 0.05 mg/kg per day for a further 2 years.
- Total: Total of all reporting groups
Arm/Group | r-hGH | Historical Control | Total
Number analyzed (Participants) | 64 | 51 | 115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 64 | 51 | 115
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 51 | 115
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Height SDS at Year 4
Description: Height SDS was calculated as height minus reference mean height divided by standard deviation of the reference population. Height SDS reflects the height relative to a reference population of the same age and gender.
Time Frame: Year 4
Population: All treated participants from r-hGH arm and all participants from Historical Control arm.
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | r-hGH | Historical Control
Number analyzed (Participants) | 61 | 51
standard deviation score | -1.35 (0.86) | -2.44 (0.73)

2. Secondary Outcome: Number of Participants With Abnormal Glycated Hemoglobin (HbA1c) Levels
Description: HbA1c develops when hemoglobin, a protein within red blood cells that carries oxygen throughout the body, joins with glucose in the blood, becoming glycated. The higher the level of glucose in the blood, the higher the level of HbA1c is detectable on red blood cells. The normal range for HbA1c is 4 percent (%) to 5.9%. Number of participants, who had abnormal HbA1c levels any time during the assessment, were reported.
Time Frame: Baseline up to Year 2
Measure: Number; unit: participants
Arm/Group | r-hGH
Number analyzed (Participants) | 61
participants | 1

3. Secondary Outcome: Difference Between Bone Age (BA) and Chronological Age (CA) (BA-CA)
Description: BA was determined using left wrist and hand X-ray. CA was determined using the date of birth. Difference of BA and CA (BA-CA) was reported.
Time Frame: Baseline, Year 1, Year 2
Population: All treated participants from r-hGH arm. This outcome measure was only planned in the r-hGH arm. Overall number of participants analyzed = participants with available data for this outcome; number analyzed = participants with available data for this outcome at specified timepoint.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | r-hGH
Number analyzed (Participants) | 60
months
  Baseline: number analyzed (Participants) | 58
  Baseline | -8.9 (7.5)
  Year 1 | -8.7 (6.5)
  Year 2: number analyzed (Participants) | 57
  Year 2 | -8.1 (7.8)

4. Secondary Outcome: Number of Participants With Anti r-hGH Antibodies
Time Frame: Baseline up to Year 2
Population: Data for this outcome was not collected from any participant.
Arm/Group | r-hGH | Historical Control
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants With Abnormal Insulin-Like Growth Factor 1 (IGF1) Levels
Description: The normal range for IGF1 levels is 45 to 117 nanogram per milliliter (ng/mL) for girls aged less than (<) 3 years and 80 to 236 ng/mL for girls aged 3 to 6 years. Values outside the normal range were considered abnormal. Number of participants, who had abnormal IGF1 levels any time during the assessment, were reported.
Time Frame: Baseline up to Year 2
Population: All treated participants from r-hGH arm. This outcome measure was only planned in the r-hGH arm.
Measure: Number; unit: participants
Arm/Group | r-hGH
Number analyzed (Participants) | 61
participants | 46

6. Secondary Outcome: Number of Participants Who Reached Normal Height at Year 4
Description: Participants with normal height were those who attained a height which was within +/- 2 height SDS of reference population standard. Height SDS was calculated as height minus reference mean height divided by standard deviation of the reference population. Height SDS reflects the height relative to a reference population of the same age and gender.
Time Frame: Year 4
Population: All treated participants from r-hGH arm. This outcome measure was only planned in the r-hGH arm.
Measure: Number; unit: participants
Arm/Group | r-hGH
Number analyzed (Participants) | 61
participants | 49

ADVERSE EVENTS:
Description: Adverse events were collected only from participants treated with r-hGH. No adverse event data collection occurred in Historical Control arm.
Arm/Group | r-hGH
Serious Adverse Events (participants affected / at risk) | 8/61
Other Adverse Events (participants affected / at risk) | 47/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | r-hGH (N=61)
Urethral reflux (Vascular disorders) | 1
Trauma leading to scalp surgery (Surgical and medical procedures) | 1
Measles (Skin and subcutaneous tissue disorders) | 1
Serious otitis (Nervous system disorders) | 1
Immunoglobulin G4 deficiency (Immune system disorders) | 1
Arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Chronic persistent cytolysis (Congenital, familial and genetic disorders) | 1
Surgery to remove large mass (meningocele/benign cyst) (Surgical and medical procedures) | 1
Transtympanic drainage tube placement (Surgical and medical procedures) | 1
Tonsillectomy/adenoidectomy (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | r-hGH (N=61)
Infection (Infections and infestations) | 47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No